CLINICAL TRIAL: NCT04974866
Title: Tyrosine Kinase Inhibitors in the Management of Local Advanced or Metastastic Adenoid Cystic Carcinoma
Brief Title: Tyrosine Kinase Inhibitors in Metastastic Adenoid Cystic Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, chief, Qingdao Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2021-07-01
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Adenoid Cystic
Keywords: Neoplasms, Glandular and Epithelial; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Neoplasms, Glandular and Epithelial; Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study drug (Experimental): EGFR TKIs
  Interventions: Drug: EGFR-TK Inhibitor

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — epidermal growth factor receptor tyrosine kinase inhibitors

SUMMARY:
There is no clinical study on epidermal growth factor receptor tyrosine kinase inhibitors has been systematically conducted in adenoid cystic carcinoma.

This is a phase II study EGFR TKIs in adenoid cystic carcinoma to evaluate its efficacy in this disease.

DETAILED DESCRIPTION:
The histologic appearance of adenoid cystic carcinoma is low grade, management of this malignancy is a challenge because of its insidious local growth pattern and lack of effency with chemotherapy or radiotherapy in metastatic disease.

In other performed clinical trials, objective responses to any cytotoxic agent or regimen are infrequent, whereas stabilization of disease was observed more commonly.

In adenoid cystic carcinoma, the study focusing on EGFR pathway is rare. According to previous study, adenoid cystic carcinoma cell lines have increased pAkt activity when EGF-stimulation is added. And when treated with EGFR/VEGFR TK dual inhibitor, the phosphorylated form of Akt decreased despite of total level of Akt is remained unchanged.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenoid cystic carcinoma
2. Local, locally-advanced or metastatic disease documented as having shown progression on a scan (CT, MRI, MIBI scan) taken 2 to 12 months prior to baseline compared to a previous scan taken at any time in the past. Progression must be documented according to RECIST criteria.
3. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent and who is previously treated with chemotherapy or local treatment (e,g transarterial chemoembolization)
4. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria
5. 18 years or older
6. ECOG performance status 0, 1, 2, 3
7. Previous treatment with chemotherapy, loco-regional therapy (e.g chemoembolization) are permitted providing that toxicity has resolved to ≤grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.
8. Adequate organ function
9. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
10. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* 1. A patient with no measurable disease, or allergy to the EGFR TKIs 2. Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry) 4. A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding 5. A pregnant or lactating patient 6. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential) 7. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study 9. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.

  10. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.

  11. Ongoing cardiac arrhythmia of grade ≥2, atrial fibrillation of any grade, or QTc interval>450msec for males or >470msec for female.

  12. A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 10 months
  progression free survival

SECONDARY OUTCOMES:
overall survival | 2 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao central Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No